CLINICAL TRIAL: NCT00955669
Title: Comparison of Autologous Transplantation of Bone Marrow Mesenchymal Stem Cells and Mononuclear Cells on Diabetic Critical Limb Ischemia and Foot Ulcer
Brief Title: Comparison of Autologous Mesenchymal Stem Cells and Mononuclear Cells on Diabetic Critical Limb Ischemia and Foot Ulcer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Department of Endocrinology and Metabolism, Southwest Hospital, Third Military Medical University, Chongqing, China, Department of Endocrinology and Metabolism, Southwest Hospital, Third Military Medical University, Chongqing, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ldb2008101
Record Dates: First submitted 2009-08-04; First posted 2009-08-10 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: Autologous Transplantation; Diabetic Foot
Keywords: mesenchymal stem cells; mononuclear cells
MeSH Terms: conditions — Diabetic Foot | interventions — Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Symptoms and Objective Examination (Active Comparator)
  Interventions: Biological: Symptoms and Objective Examination

INTERVENTIONS:
Biological: Symptoms and Objective Examination — 5.0*108~5.0*109 MSCs and MNCs were transplant into impaired lower limbs by intramuscular injection
  Other Names: transplant

SUMMARY:
Objective:

To compare the effect and safety of autologous transplantation of bone marrow mesenchymal stem cells(MSCs) and mononuclear cells(MNCs) on Diabetic patients with Critical Limb Ischemia and Foot Ulcer.

Methods:

patients were randomized into the A group and the B group by use of a randomization table. One lower limb in A group or in B group was selected randomly for MSCs or MNCs transplantation as MSCs or MNCs group, the other lower limb in the same patient was selected for placebo（normal saline ,NS）injection as NS group.

The whole procedures of this clinical trial were blinded to both patients and investigators.Patients in both groups received the same ordinary treatment. Meanwhile, MSCs and MNCs were transplanted into the impaired lower limbs respectively. Follow-up index include: efficacy (pain,ulcer healing rate, lower limb amputation rate and ,ankle-brachial index,Transcutaneous oxygen pressure,magnetic resonance angiography) and safety (infection of the injection site, immunological rejection, and tumour generation).

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS Written informed consent was obtained from all subjects. Type 2 diabetic patients with bilateral critical limb ischemia (ankle-brachial index, ABI from 0.30 to 0.60) and at least with one foot ulcer, but without malignant tumor or gangrene above the ankle and/or severe coronary, cerebral and renal vascular disease, were eligible for the participation in this trial. Eligible patients took part in this study on a voluntary basis. They were randomized into the A and B group by use of a randomization table. One lower limb in A group or in B group was selected randomly for BMMSCs or BMMNCs transplantation as BMMSCs or BMMNCs group, the other lower limb in the same patient was selected for placebo（normal saline ,NS）injection as NS group. The whole procedures of this clinical trial were blinded to both patients and investigators.

Preparation of Human Autologous Serum Preparation of MSCs and MNCs Flow Cytometric Analysis Examination of cells Safety Administration of therapy 5.0*108~5.0*109 MSCs and MNCs were transplant into impaired lower limbs by intramuscular injection.

observation index and assessment guidelines Statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Age from 40 to 70 years
* Type 2 diabetic patients
* bilateral critical limb ischemia(ABI from 0.30 to 0.60)
* at least with one foot ulcer

Exclusion Criteria:

* dry gangrene above the ankle or moist gangrene
* malignant tumor
* severe coronary,cerebral and renal vascular disease

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Magnetic resonance angiography | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chen bing, doctor, Study Director — Endocrinology and Metabolism Department, the south west Hospital of the Third Military Medical University
Locations (1):
- the southwest Hospital, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Lu D, Jiang Y, Deng W, Zhang Y, Liang Z, Wu Q, Jiang X, Zhang L, Gao F, Cao Y, Chen B, Xue Y. Long-Term Outcomes of BMMSC Compared with BMMNC for Treatment of Critical Limb Ischemia and Foot Ulcer in Patients with Diabetes. Cell Transplant. 2019 May;28(5):645-652. doi: 10.1177/0963689719835177. Epub 2019 Mar 27. PMID 30917698
- [Derived] Chen Y, Ma Y, Li N, Wang H, Chen B, Liang Z, Ren R, Lu D, Boey J, Armstrong DG, Deng W. Efficacy and long-term longitudinal follow-up of bone marrow mesenchymal cell transplantation therapy in a diabetic patient with recurrent lower limb bullosis diabeticorum. Stem Cell Res Ther. 2018 Apr 10;9(1):99. doi: 10.1186/s13287-018-0854-9. PMID 29631615